CLINICAL TRIAL: NCT00584844
Title: A Longitudinal Phase 2 Study for the Continued Evaluation of the Safety and Immunogenicity of a Live Francisella Tularensis Vaccine, NDBR 101, Lot 4
Brief Title: Safety and Immunogenicity Study of a Live Francisella Tularensis Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: A-12775; FY03-24 (Other: SIP)
Record Dates: First submitted 2007-12-20; First posted 2008-01-02 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Tularemia
Keywords: Live Vaccine Strain (LVS), Bacterial Infections, Ulceroglandular, Oculoglandular
MeSH Terms: conditions — Tularemia; Bacterial Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- F tularensis Vaccine (0.0025 mL) (Experimental): Subjects receive a small amount of F tularensis vaccine (0.0025mL) placed on a cleansed site on the skin on the volar surface of the forearm. A bifurcated needle was used to make 15 superficial punctures at the vaccination site to permit percutaneous penetration of the vaccine.
  Interventions: Biological: Live F tularensis Vaccine

INTERVENTIONS:
Biological: Live F tularensis Vaccine — Subjects will receive one drop of reconstituted F tularensis vaccine (approximately 0.0025 ml), applied with a bifurcated needle to the volar surface of the forearm, and the skin will be pricked 15 times over the prepared area. A booster dose will be given at the same dose volume and route of administration if the titer (days 56-84) is inadequate (< 1:20).

SUMMARY:
This study is designed to determine the safety and immunogenicity of a Live Francisella tularensis Vaccine

DETAILED DESCRIPTION:
Study was designed as a continuation of previously published research and targets subjects who were at risk of occupational exposure to F tularensis virus. Based on screening examinations; if a subject had a positive baseline titer (<1:20) and gave no history of significant exposure to F tularensis or history of tularemia disease, had never received tularemia vaccination, and was at risk of exposure to F tularensis they could be enrolled in this protocol to receive vaccination. Subjects returned for follow-up exams on Days 1, 2, and 7; once between Days 12 and 16; and once between Days 28 and 35 post-vaccination. If titers; after blood samples on Days 28, 35 and 12 months showed <1:20 the vaccination could be repeated at Days 56-84. If the repeat titer remained <1:20, a booster vaccination could be administered. Subjects could be boosted 2 times with 1 year. If the titer measured 12 months after vaccination (+30 days) was >1:20 and the subject had no lingering AEs, the subjects participation was considered complete.

ELIGIBILITY:
Inclusion Criteria:>

* At least 18 years old, or if on active military duty, 17 years old >
* Females of childbearing potential must agree to have a urine pregnancy test immediately before vaccination (Exception: documented hysterectomy or > 3 years of menopause). The results must be negative. Volunteers must agree not to become pregnant for 3 months after receipt of the vaccine.>
* Subject must be actively enrolled in the SIP >
* Subjects must be considered at risk for exposure to F. tularensis.>
* Subjects must have an up-to-date (within 1 year) medical history, physical examination, and laboratory tests on their charts and be medically cleared for participation by an investigator. Examinations or tests may be repeated within 1 year at the discretion of the enrolling physician.>
* Volunteer must be willing to return for all follow-up visits on days 1, 2, 7, once between days 12-16, and once between days 28-35, days 56-84 (if needed), all visits for serology, as well as an annual visit while enrolled in protocol.>
* Volunteer must agree to report any Adverse Event which may or may not be associated with administration of the test article for at least 28 days after vaccination. All Serious and Unexpected Adverse Events will be reported for the duration of the volunteer's participation in the study. >

Exclusion Criteria:>

* Clinically significant abnormal lab results including evidence of Hepatitis C*, Hepatitis B* carrier state, or elevated liver function tests (2X normal values or at discretion of PI).>
* Personal history of an immunodeficiency or current treatment with an oral or intravenous immunosuppressive medication.>
* Confirmed HIV* infection.>
* Any other medical condition at the discretion of the PI.>
* Antibiotic therapy for 7 days before vaccination.>
* Females must not be pregnant or lactating (females must agree to not become pregnant for 3 months after vaccination).>
* Any known allergies to excipients of the vaccine>
* Administration of another live vaccine within 4 weeks or an inactivated vaccine (generally) within 7 days of tularemia vaccination.>
* Any unresolved adverse event resulting from a previous immunization. >

Ages: 17 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 484 (Actual)
Dates: Start 2004-10; Primary Completion 2009-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Goldberg, MD, Principal Investigator — USAMRIID Medical Division
Locations (1):
- U.S. Army Medical Research Institute of Infectious Diseases, Fort Deterick, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment at the Special Immunizations Clinic at USAMRIID is expected to last 5 years and include up to 1,000 subjects who were at risk of occupational exposure to F tularensis.
Period: Overall Study
Arm/Group | F Tularensis Vaccine (0.0025 mL)
Started | 484
Completed | 405
Not Completed | 79
Not completed — Withdrawal by Subject | 59
Not completed — Screen Failure | 20

BASELINE CHARACTERISTICS:
Arm/Group | F Tularensis Vaccine (0.0025 mL)
Number analyzed (Participants) | 405
Age, Customized [Count of Participants; unit: Participants]
  <20 years | 2
  20-29 years | 108
  30-39 years | 126
  40-49 years | 106
  50-59 years | 54
  60-69 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145
  Male | 260
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23
  Not Hispanic or Latino | 382
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 13
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 20
  White | 357
  More than one race | 11
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 405

OUTCOME MEASURES:

1. Primary Outcome: Safety: Adverse Event Category Rates for All Vaccinations
Description: AE analysis was conducted for all intent-to-treat subjects regardless of compliance with titer schedule.
Time Frame: AEs/SAEs recorded through duration of study; immunogenicity via MA on days 0, 28-35, 56-84, and at 1 year
Measure: Number; unit: Adverse events
Groups:
- Males: All males in study
- Females: All females in study
Arm/Group | Males | Females
Number analyzed (Participants) | 294 | 168
Adverse events
  Any AE: Mild | 264 | 162
  Any AE: Moderate | 53 | 48
  Any AE: Severe | 11 | 10
  Local: Mild | 248 | 153
  Local: Moderate | 7 | 13
  Locale: Severe | 0 | 1
  Systemic: Mild | 121 | 105
  Systemic: Moderate | 48 | 42
  Systemic: Severe | 11 | 9
  Relationship: Unrelated | 30 | 28
  Relationship: Unlikely | 33 | 29
  Relationship: Possible | 86 | 77
  Relationship: Probable | 62 | 41
  Relationship: Definate | 246 | 153
  Outcome: Resolved | 271 | 163
  Outcome: Resolved with sequelae | 4 | 1
  Treatment required:None | 260 | 160
  Treatment required: Intervention required | 75 | 75
  Treatment required: Other | 7 | 1
  Treatment required: Hospitalization | 6 | 6

2. Secondary Outcome: Immunogenicity: Protocol Compliant Post-primary Titer Rates
Description: Percentage of subjects with less than or greater than titers (> or < 1:20) for compliant post-primary titers.
Time Frame: 12 months
Population: As stated in the protocol, only titers taken in compliance with the prescribed schedule were used in the statistical analysis. 454 were compliant and analyzed.
Measure: Number; unit: Percentage of subjects
Groups:
- Percent of Subjects: Percentage of subjects in specific category
Arm/Group | Percent of Subjects
Number analyzed (Participants) | 454
Percentage of subjects
  Days 28-35: All subjects <1.20 | 4.1
  Days 28-35: All subjects >1.20 | 95.9
  Days 56-84: All subjects <1.20 | 73.3
  Days 56-84: All subjects >1:20 | 26.7
  Month 12: All subjects <1:20 | 3.6
  Month 12: All subjects >1:20 | 96.4
  Overall: <1:20 | 2.6
  Overall: >1:20 | 97.4

3. Secondary Outcome: Immunogenicity: Protocol-compliant Post-boost 1 Titer Rates
Description: Percentage of subjects with less than or greater than titers (> or < 1:20) who received post-boost 1
Time Frame: 12 months
Population: As stated in the protocol, only titers taken in compliance with the prescribed schedule were used in the statistical analysis. 19 were compliant and analyzed.
Measure: Number; unit: Percentage of subjects
Arm/Group | Percent of Subjects
Number analyzed (Participants) | 19
Percentage of subjects
  Days 28-35: <1:20 | 22.2
  Days 28-35: >1:20 | 77.8
  Days 56-84: <1:20 | 100.0
  Days 56-84: >1:20 | 0
  Month 12: <1:20 | 43.8
  Month 12: >1:20 | 56.3
  Overall: <1:20 | 26.3
  Overall: >1:20 | 73.7

4. Secondary Outcome: Immunogenicity: Protocol-compliant Post-boost 2 Titer
Description: Percentage of subjects with less than or greater than titers who received post-boost 2.
  Responder = > 1:20 Non-responder = < 1:20
Time Frame: 12 months
Population: As stated in the protocol, only titers taken in compliance with the prescribed schedule were used in the statistical analysis. 18 were compliant and analyzed.
Measure: Number; unit: Percentage of subjects
Arm/Group | Percent of Subjects
Number analyzed (Participants) | 18
Percentage of subjects
  Days 28-35: Non-Responder | 5.6
  Days 28-35:Responder | 94.4
  Days 56-84: Non-Responder | 25.0
  Days 56-84: Responder | 75.0
  Month 12: Non-Responder | 6.3
  Month 12: Responder | 93.8
  Overall: Non-Responder | 5.3
  Overall: Responder | 94.7

ADVERSE EVENTS:
Time Frame: 12 months
Description: AE analysis was conducted for all intent-to-treat subjects regardless of compliance with titer schedule. A single AE greater than 1 day duration that changed in severity was tabulated as one AE with only the highest severity coding. AE's were assessed on Days 1, 2, 7, 12-16, 28-35, 56-84 and 12 months.
Groups:
- Mild: Mild
- Moderate: Moderate
- Severe: Severe
Arm/Group | Mild | Moderate | Severe
Serious Adverse Events (participants affected / at risk) | 0/462 | 10/462 | 11/462
Other Adverse Events (participants affected / at risk) | 426/462 | 101/462 | 21/462
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mild (N=462) | Moderate (N=462) | Severe (N=462)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Malaria (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pilonidal cyst (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Meniscus lesion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Spondylolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mild (N=462) | Moderate (N=462) | Severe (N=462)
Lymph node pain (Blood and lymphatic system disorders) | 17 (17) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 79 (82) | 2 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ear congestion (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 2 (2) | 3 (3) | 0 (0)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eye discharge (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 2 (2) | 2 (2) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Aphthous stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 10 (10) | 3 (3) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 18 (18) | 8 (8) | 2 (2)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Axillary pain (General disorders) | 79 (79) | 6 (6) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 6 (7) | 5 (5) | 0 (0)
Fatigue (General disorders) | 36 (36) | 11 (11) | 2 (2)
Feeling hot (General disorders) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site discharge (General disorders) | 2 (2) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 355 (370) | 8 (8) | 1 (1)
Injection site exfoliation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site induration (General disorders) | 104 (104) | 0 (0) | 0 (0)
Injection site oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 79 (79) | 2 (2) | 0 (0)
Injection site paraesthesia (General disorders) | 3 (3) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 111 (111) | 1 (1) | 0 (0)
Injection site rash (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site vesicles (General disorders) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 40 (40) | 9 (9) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pain (General disorders) | 14 (14) | 3 (3) | 1 (1)
Pyrexia (General disorders) | 12 (12) | 8 (8) | 1 (1)
Vaccination site pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Injection site pustule (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lymphangitis (Infections and infestations) | 4 (4) | 0 (0) | 0 (0)
Malaria (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pilonidal cyst (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 6 (6) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Animal scratch (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Eye injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Limb crushing injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Meniscus lesion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 6 (6) | 0 (0) | 0 (0)
Lymph node palpable (Investigations) | 19 (19) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 30 (34) | 4 (4) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 1 (1)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 17 (19) | 3 (4) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 6 (6) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 23 (23) | 5 (5) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 0 (0) | 1 (1)
Nodule on extremity (Musculoskeletal and connective tissue disorders) | 10 (10) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 42 (43) | 5 (5) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Spondylolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 7 (7) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 86 (86) | 23 (23) | 3 (3)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Sinus headache (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0)
Tension headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Bladder discomfort (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 23 (23) | 3 (3) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 27 (27) | 5 (5) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 34 (34) | 6 (6) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 3 (3) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 0 (0) | 0 (0)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus operation (Surgical and medical procedures) | 3 (3) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No